CLINICAL TRIAL: NCT06889272
Title: Investigation of the Relationship Between Blood Transfusion Volume and Development of Renal Failure in Pediatric Patients Undergoing Cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Murat İzgi, Assistant Professor, Hacettepe University
Other Study IDs: Yusuf CELIK; Murat IZGI (Other: Hacettepe Univercity)
Record Dates: First submitted 2025-02-18; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Congenital Cardiac Defect; Acute Renal Injury; Blood Transfusion Complication
MeSH Terms: conditions — Heart Defects, Congenital; Acute Kidney Injury; Transfusion Reaction | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with acute kidney injury: blood transfusion during surgery
  Interventions: Other: blood transfusion
- patients without acute kidney injury: blood transfusion during surgery
  Interventions: Other: blood transfusion

INTERVENTIONS:
Other: blood transfusion — Red blood cell suspension replacement during surgery

SUMMARY:
Blood transfusion strategies in cardiac surgery are a research topic that has been studied more for adults. There is not enough data on this subject for children in studies. Investigators aim to examine the renal damage risk level of blood transfusion volume, which is one of the modifiable risk factors that can cause acute kidney injury in pediatric cases undergoing cardiac surgery.

The main question it aims to answer is:

What is the effect of blood transfusion volume on the risk of renal damage in pediatric cardiovascular surgery? The names of the patients who were operated on by the Department of Cardiovascular Surgery will be accessed from the system records and their files will be reviewed. The patients' demographic information, anesthesia management and postoperative renal function tests will be scanned.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing cardiovascular surgery

Exclusion Criteria:

* Being over 18 years old Weighting over 30 kg Preoperative acute kidney injury

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients who applied to Hacettepe University Faculty of Medicine (HÜTF) Hospital and underwent cardiac surgery by the Department of Cardiovascular Surgery between January 1, 2013 and December 31, 2023 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
postoperative acute renal failure | From registration to the end of the second postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Murat Izgi, Study Director — Assistant professor
Locations (1):
- Hacettepe University Anesthesiology and Reanimation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided